CLINICAL TRIAL: NCT04060017
Title: Early Treatment of Language Impairment in Young Children With Autism Spectrum Disorder With Leucovorin Calcium
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: State University of New York - Downstate Medical Center (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Frye, Principal Investigator, Southwest Autism Research & Resource Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOD Leucovorin
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Language Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Language Disorders | interventions — Leucovorin

STUDY DESIGN:
Intervention Model Description: Prospective randomized 12-week double-blind placebo-controlled study followed by 12-week open label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple masking during blinded phase, followed by unblinding during open label phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-leucovorin calcium (Experimental): The liquid form of leucovorin calcium will be dosed by weight, with a target dose of 1mg/kg/day, divided into two daily doses. This product may be taken alone or mixed with liquid. Participants randomized to this arm will receive active treatment for both 12-week phases of the study.
  Interventions: Drug: Levoleucovorin Calcium
- Placebo (Placebo Comparator): The placebo will mimic the experimental treatment in flavor, odor, packaging, and dosing instructions. Participants randomized to this arm will receive placebo for the first 12 weeks of the study, then active treatment for the remaining 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levoleucovorin Calcium — Liquid leucovorin calcium dosed by weight
  Other Names: L-leucovorin; L-leucovorin calcium; L-folinic acid, calcium salt; L-folinate, calcium salt
  Arms: L-leucovorin calcium
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the cognitive and behavioral effects of liquid leucovorin calcium on young children with autism spectrum disorder (ASD) and determine whether it improves language as well as the core and associated symptoms of ASD. The investigators will enroll 80 children across two sites, between the ages of 2.5 and 5 years, with confirmed ASD and known language delays or impairments. Participation will last approximately 26 weeks from screening to end of treatment.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder with life-long consequences that affects young children during critical times in their development. ASD is defined by impairments in social-communication as well as the presence of restricted interests and repetitive behaviors. ASD is frequently associated with co-occurring language delays. Currently the only well-accepted treatment for core ASD symptoms is behavior therapy such as Applied Behavioral Analysis and Early Intensive Behavioral Intervention. There is no US Food and Drug Administration approved medical therapy that addresses core ASD symptoms or the pathophysiological processes that underlie ASD.

The primary aim of this study is to evaluate the effect of a liquid form of leucovorin calcium on language impairments in very young children with ASD. Participants entered into the trial will have delayed social and communication abilities known to be associated with ASD. The investigators hypothesize that leucovorin calcium will significantly improve language as well as core and associated behavioral symptoms of ASD, and be well-tolerated with no significant adverse effects, in young children with ASD. The investigators further hypothesize that a combination of baseline cellular and genetic biomarkers will predict cognitive and behavioral response to the intervention.

To assess whether the liquid form of leucovorin calcium is superior to placebo, the investigators will study 80 children across two sites, between the ages of 2.5 and 5 years, with confirmed ASD and known language delays at baseline. Participants will be randomly assigned to receive active treatment or placebo for 12 weeks under double-blind conditions. At the end of 12 weeks, all participants will receive active treatment for 12 weeks. Language skills, as well as specimen biomarkers, will be measured at screening and after each treatment arm in order to determine if the supplement positively influences language ability.

ELIGIBILITY:
Inclusion Criteria:

1. Autism Spectrum Disorder (as defined below).
2. Between 2 years 6 months and 5 years 2 months of age at baseline
3. Language impairment (Ages and Stage Questionnaire between -1 and -3 SD for Language)
4. Has at least 4 month old expressive language ability as assessed by the MSEL Expressive Language Scale (i.e., Parent answers "yes" to " Voluntary babbling (such as 'bu, bu, bu")" Question #7 on the MSEL Expressive Language Scale.
5. English included in the languages in which the child is being raised
6. Autism severity of moderate or higher (≥4) under the 7-item clinical global impression-severity scale. Moderate level of autism severity (4) is defined by the diagnosis of ASD with language impairment, so fulfilling #1 and #4 fulfills this requirement.

6. Ability to maintain all ongoing complementary, dietary, traditional, and behavioral treatments constant for the study period 7. Unchanged complementary, dietary, traditional, and behavioral treatments for two months prior to study entry

Exclusion Criteria:

1. Known FRAA status by clinically validated test performed outside of research studies.
2. Mineral or vitamin supplementation that exceeds the Tolerable Upper Daily Intake Levels set by the Institute of Medicine (See Table 5 below)
3. Significant self-abusive or violent behavior or evidence of suicidal ideation, plan or behavior
4. Severely affected as defined by CGI-Severity Standard Score = 7 (Extremely Ill)
5. Severe prematurity (<34 weeks gestation) as determined by medical history
6. Current uncontrolled gastroesophageal reflux
7. Current or history of liver or kidney disease as determined by medical history and safety labs
8. Genetic syndromes
9. Congenital brain malformations
10. Epilepsy
11. Any medical condition that the PI determines could jeopardize the safety of the study subject or compromise the integrity of the data
12. Significant negative reaction (i.e. fainting, vomiting, etc.) because of a previous blood draw.
13. Failure to thrive or Body Mass Index < 5%ile or <5%ile for weight (male <11.2kg; female <10.8kg by CDC 2000 growth charts) at the time of screening.
14. Concurrent treatment with drug that would significantly interact with l-leucovorin such as specific chemotherapy agents, antimalarial and immune suppressive agents and select antibiotics (See Table 6 below).
15. Allergy or Sensitivity to ingredients in the investigational product or placebo
16. Evaluation with the MSEL or BOSCC within 3 months of entering the study
17. Planned evaluation with the MSEL or BOSCC during the study

Ages: 30 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in measures of expressive language | Screening, Week 12, Week 24
  Mullen Scales of Early Learning: a scale of cognitive abilities across the following domains: gross motor (not a core subscale), visual reception, fine motor, expressive language, and receptive language. Total change in expressive language ability will be measured by the change in the expressive language raw score. The expressive language domain is a 28-item scale with a raw score range of 0-50. Changes in expressive language raw scores will be reported. A higher raw score indicates a higher level of language ability.

SECONDARY OUTCOMES:
Evaluate the change in measures of receptive language | Screening, Week 12, Week 24
  Mullen Scales of Early Learning: a scale of cognitive abilities across the following domains: gross motor (not a core subscale), visual reception, fine motor, expressive language, and receptive language. Total change in receptive language ability will be measured by the change in the receptive language raw and t score. The receptive language domain is a 33-item scale with a raw score range of 0-48 and a t score range of 20-80. T scores are calculated from the raw score and based on age norms. Changes in receptive language raw and t scores will be reported. A higher raw and t score indicates a higher level of language ability. In addition, we will analyze change in expressive language t-score.
Evaluate the safety and tolerability of L-leucovorin calcium in young children with ASD | Screening, Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 24
  Modified Dosage Record and Treatment Emergent Symptoms: treating clinician will perform a review of medical and behavioral history at each visit to assess incidence of treatment-emergent adverse events. The treating clinician will use the scale to record presence and intensity of adverse effects. Intensity is rated on a scale of 0 (Not present) to 3 (Severe). The treating clinician will also judge the adverse effects' relatedness to treatment. Relatedness is rated on a scale of 1 (None) to 4 (Defined). The treating clinician will denote action taken. Action taken is rated on a scale of 0 (None) to 5 (Discontinue Treatment). No total score is calculated. However, higher ratings on any individual item indicate greater severity of adverse effects.
Evaluate the safety of L-leucovorin calcium in young children with ASD | Screening, Week 12, Week 24
  Routine comprehensive blood panels will be collected to determine whether treatment-emergent basic blood chemistry is altered. Presence of any changes during the course of study enrollment will be evaluated by the treating physician and determined clinically significant or not clinically significant. If determined by the treating physician, a change will be considered an adverse event.
Evaluate the safety of L-leucovorin calcium in young children with ASD on antiepileptic drugs | Screening, Week 12, Week 24
  For children using antiepileptic drugs, the level of that drug will be measured. If determined by the treating physician, a change will be considered an adverse event.
Evaluate the overall change in core autism symptoms of social communication | Screening, Week 12, Week 24
  Brief Observation of Social Communication Change: a 16-item scale that rates social interactions between children with ASD and their interactive rater. Each item is rated on a scale of 0-5, wherein 0 indicates the least severe behavior and 5 indicates the most severe behavior. A higher score is indicative of more severe social communication deficits. Because this evaluation is not valid with PPE it will not be performed during evaluation when PPE is required
Evaluate the change in stereotypical autism symptoms | Screening, Week 6, Week 12, Week 24
  Aberrant Behavior Checklist-2: a 58-item parent-reported measure of stereotypical autism behaviors with ratings in the following domains: irritability, social withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech. Each item is rated from 0 (Not a Problem) to 3 (Severe Problem). The raw score will be reported. The total raw score is the sum of the domain raw scores. A higher raw score in any of the domains indicates more severe problems in that domain; a higher total raw score indicates more severity of stereotypical autism symptoms overall.
Evaluate the change in social withdrawal autism symptoms | Screening, Week 6, Week 12, Week 24
  Aberrant Behavior Checklist-2: a 58-item parent-reported measure of stereotypical autism behaviors with ratings in the following domains: irritability, social withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech. Each item is rated from 0 (Not a Problem) to 3 (Severe Problem). The raw score will be reported. The total raw score is the sum of the domain raw scores. A higher raw score in any of the domains indicates more severe problems in that domain; a higher total raw score indicates more severity of stereotypical autism symptoms overall.
Evaluate the change in effects of autism symptoms most problematic to family members | Screening, Week 6, Week 12, Week 24
  Parent Target Problems: a parent-nominated list of 2 most problematic core autism symptoms. Responses are documented in a brief narrative and detail frequency, constancy, intensity, and impact of behavior on the family. Subjective reports of frequency, constancy, intensity, and impact on family will be rated by a blinded statistician at the conclusion of the study. Higher scores indicate more severe impact on family.
Evaluate change in overall autism severity | Baseline, Week 6, Week 12, Week 24
  Clinical Global Impression Scale: The Clinical Global Impression Scale-Severity is a 7-point measure of overall symptom severity, ranging from 1 (Normal) to 7 (Extreme), with a raw score range of 1-7. The raw score will be reported. The Clinical Global Impression Scale-Improvement is a measure in change of symptom severity, ranging from 1 (Very Much Improved) to 7 (Very Much Worse). A Score of 4 indicates no change in symptom severity.
Evaluate change in autism severity of specific symptoms | Baseline, Week 6, Week 12, Week 24
  Ohio State University Clinical Impressions Scale: a clinical rating of severity and improvement of 10 autism domains: social interaction, aberrant/abnormal behavior, repetitive/ritualistic behavior, verbal communication, non-verbal communication, hyperactivity/inattention, anxiety/fears, sensory sensitivities, restricted/narrow interests, autism. Severity will be measured at baseline. Each item is rated from 1 (Normal) to 7 (Among the most severe) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment. At the following time points, improvement will be measured. Each item is rated from 1 (Very much improved) to 7 (Very much worse) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment.
Evaluate the change in overall cognitive ability | Baseline, Week 12, Week 24
  Mullen Scales of Early Learning: a scale of cognitive abilities across core domains: visual reception, fine motor, expressive language, receptive language. Expressive language domain: 28-item scale with a raw score range of 0-50, t score range of 20-80. Receptive language domain: 33-item scale with a raw score range of 0-48, t score range of 20-80. Visual reception domain: 33-item scale with a raw score range of 0-50, t score range of 20-80. Fine motor domain: 33-item scale with a raw score range of 0-50, t score range of 20-80.
  Change in domain ability will be measured by the change in domain t score. T scores are calculated from raw scores and based on age norms. A higher domain t score indicates a higher level of ability in that domain. Domain t scores will be used to get a standard composite score. Change in cognition will be measured by change in the Early Learning Composite standardized Scaled score. A higher composite score indicates higher overall cognitive ability.
Evaluate the change in adaptive functioning | Baseline, Week 12, Week 24
  Vineland Adaptive Behavior Scale-II Domain LevelI: a scale to assess adaptive behavior in children with developmental/intellectual disabilities. This is a 135-item parent-reported measure with ratings in the following domains: communication, daily living skills, and socialization. The frequency of each item is scaled from 0 (Never) to 2 (Usually). For each domain, there are 45 items with a maximum score of 90. Change in each domain will be measured by the change in standard score. Standard scores are calculated from the raw scores and based on age norms. A higher standard score in any domain indicates a higher level of adaptive behavior in that domain. Domain standard scores will be used to get a standard composite score. Change in adaptive behavior will be measured by the change in the standard score. A higher composite score indicates higher overall adaptive behavior ability.
Evaluate the change in social withdrawal autism symptoms | Baseline, Week 6, Week 12, Week 24
  Social Responsiveness Scale Preschool Version. The Social Responsiveness Scale is a quantitative scale that measures severity and type of social impairments that characterize ASD. It is a standard measure in ASD clinical trials. We will use the preschool version to match the age range of our study.

OTHER OUTCOMES:
Test if biomarkers (FRAAs) predict clinical response to L-leucovorin | Screening
  FRAA titers (described above) will be measured and analyzed as a predictive variable in treatment outcomes.
Test if biomarkers (single nucleotide polymorphisms) predict clinical response to L-leucovorin | Screening, Week 12
  Saliva will be collected to determine presence of the following single nucleotide polymorphisms: MTR, MTHFR6, DHFR, GCH1, MTHFR12, RFC, FOLH, COMT. Presence or absence of these genetic polymorphisms will be analyzed to assess correlation with response to L-leucovorin treatment.
Combine presence of FRAA titers and single nucleotide polymorphisms (above) into a predicting equation that will evaluate the probability of positive response to L-leucovorin treatment. | Up to 1 year after study completion
  A combination of FRAA titers and single nucleotide polymorphisms will be analyzed along with outcome data to predict response to L-leucovorin. Presence or absence of one or both of these biomarkers will be analyzed to assess how these biomarkers correlate with treatment outcome (i.e. whether the treatment was effective).

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Principal Investigator — Rossignol Medical Center
Locations (2):
- United States (2):
  - Southwestern Autism Research & Resource Center, Phoenix, Arizona
  - State University of New York, Downstate, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No
The investigators plan to publish the results of the study in an academic journal. Results may also be shared at conferences and presentations.

REFERENCES:
- [Background] Frye RE, Sequeira JM, Quadros EV, James SJ, Rossignol DA. Cerebral folate receptor autoantibodies in autism spectrum disorder. Mol Psychiatry. 2013 Mar;18(3):369-81. doi: 10.1038/mp.2011.175. Epub 2012 Jan 10. PMID 22230883
- [Background] Frye RE, Rossignol DA, Scahill L, McDougle CJ, Huberman H, Quadros EV. Treatment of Folate Metabolism Abnormalities in Autism Spectrum Disorder. Semin Pediatr Neurol. 2020 Oct;35:100835. doi: 10.1016/j.spen.2020.100835. Epub 2020 Jun 25. PMID 32892962
- [Background] Frye RE, Slattery JC, Quadros EV. Folate metabolism abnormalities in autism: potential biomarkers. Biomark Med. 2017 Aug;11(8):687-699. doi: 10.2217/bmm-2017-0109. Epub 2017 Aug 3. PMID 28770615
- [Background] Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, Sailey A, Wynne R, Rose S, Melnyk S, Jill James S, Sequeira JM, Quadros EV. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Mol Psychiatry. 2018 Feb;23(2):247-256. doi: 10.1038/mp.2016.168. Epub 2016 Oct 18. PMID 27752075
- [Background] Frye RE, Delhey L, Slattery J, Tippett M, Wynne R, Rose S, Kahler SG, Bennuri SC, Melnyk S, Sequeira JM, Quadros E. Blocking and Binding Folate Receptor Alpha Autoantibodies Identify Novel Autism Spectrum Disorder Subgroups. Front Neurosci. 2016 Mar 9;10:80. doi: 10.3389/fnins.2016.00080. eCollection 2016. PMID 27013943